CLINICAL TRIAL: NCT00810069
Title: Comparison of Two Different Treatment Strategies in Patients With Major Depressive Disorder Not Exhibiting Improvement on Escitalopram Treatment: Early vs. Delayed Intervention Strategy
Brief Title: Early Versus Delayed Switch in Medication in Patients With Major Depressive Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli LIlly
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12329; F1J-EW-HMGD (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-12-16; First posted 2008-12-17 (Estimated); Results first posted 2011-06-21 (Estimated); Last update posted 2011-06-21 (Estimated); Status verified 2011-05

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; MDD; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Duloxetine Hydrochloride; Escitalopram; Dexetimide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early Intervention (Experimental): Escitalopram 10 milligrams per day for 4 weeks (one 10 milligram [mg]-capsule) followed by Duloxetine flexible dose (60 or 120 mg daily) for 12 weeks.
  Interventions: Drug: Duloxetine Hydrochloride; Drug: Escitalopram
- Delayed Intervention (Experimental): Escitalopram 10 mg per day for 4 weeks (one 10 mg-capsule) followed by Escitalopram 10 to 20 mg per day for 4 weeks (one or two 10 mg capsule[s]). Then, non-responders switched to Duloxetine 60 or 120 mg per day for 8 weeks , and responders continued on Escitalopram 10 to 20 mg per day for 8 weeks.
  Interventions: Drug: Duloxetine Hydrochloride; Drug: Escitalopram

INTERVENTIONS:
Drug: Duloxetine Hydrochloride — Flexible dose of 60 or 120 mg daily
  Other Names: Cymbalta; LY248686
Drug: Escitalopram — 10 mg in both Early and Delayed Intervention. Flexible dose of 10 to 20 mg daily in Delayed Intervention.
  Other Names: Lexapro; Cipralex

SUMMARY:
This study investigates two different approaches to the change in antidepressant treatment when an initial treatment is not effective: early intervention or delayed intervention.

Two hypothesis will be tested:

1. that time to confirmed response is shorter in the early intervention strategy vs. delayed intervention strategy
2. that the time to confirmed remission is shorter in the early intervention strategy compared to delayed intervention strategy.

ELIGIBILITY:
Inclusion Criteria

1. Male or female participants of at least 18 years of age who meet criteria for Major Depressive Disorder (MDD), single or recurrent episode according to the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV®-TR) disease diagnostic criteria.
2. Participants (receiving or not antidepressant treatment) who, based on investigator criteria, initiate treatment with escitalopram or change their current Alzheimer's Disease (AD) treatment to escitalopram for this current MDD episode, at the initial visit.
3. Must have a baseline score of ≥ 19 on the 17-item Hamilton Depression Rating Scale (HAMD-17) at the initial visit.
4. Must have a baseline score of ≥ 4 in the Clinical Global Impression-Severity Scale (CGI-S) at the initial visit.
5. Have a level of understanding sufficient to provide Informed Consent Document (ICD), and to communicate with the investigators and site personnel.
6. Are judged to be reliable and agree to keep all appointments for clinic visits and procedures required by the protocol.

   Exclusion Criteria:
7. Have any current primary Axis I disorder other than MDD, including but not limited to dysthymia.
8. Have a diagnosis of dementia, Alzheimer's disease (AD), or organic brain syndrome; or who are cognitively impaired or who have language problems that prevent them from understanding and/or providing valid answers to the rating scale contents.
9. Concomitant participation in other studies with investigational or marketed products.
10. Are not expected to be able to be monitored throughout the entire study period for reasons unrelated to their illness (for instance, change of residence or healthcare center of reference).
11. Are demonstrating a response or demonstrated a response to the AD treatment for the current depression episode previous to baseline visit.
12. Are investigator site personnel directly affiliated with this study and/or their immediate families. "Immediate family" is defined as a spouse, parent, child, or sibling, whether biological or legally adopted.
13. Are employed by Lilly or Boehringer Ingelheim (BI) (that is, employees, temporary contract workers, or designees responsible for the conduct of the study). Immediate family of Lilly or BI employees may participate in Lilly or BI-sponsored clinical trials, but are not permitted to participate at a Lilly or BI facility. "Immediate family" is defined as a spouse, parent, child, or sibling, whether biological or legally adopted.
14. Women of childbearing potential who are not using a medically accepted means of contraception (for example, intrauterine device, oral contraceptive, contraceptive patch, implant, Depo-Provera [medroxyprogesterone acetate injectable suspension, Pharmacia & Upjohn], or barrier devices) when engaging in sexual intercourse. Women who are pregnant or breast-feeding may not participate in the study.
15. Have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry.
16. Are judged to be at serious suicidal risk in the opinion of the investigator, and/or if the participant's baseline (Visit 1) HAMD-17 scores on item 3 suicide are 3.
17. Have been treated with a monoamine oxidase inhibitor (MAOI) within 14 days prior to Visit 1 or potential need to use an MAOI during the study or within 5 days after discontinuation of study drug.
18. Require initiation or discontinuation of psychotherapy within 6 weeks prior to enrollment (Visit 1) or at any time during the study.
19. Have any contraindication for the use of duloxetine based on Duloxetine Summary of Product Characteristics (SPC) or any contraindication for the use of escitalopram based on Escitalopram SPC.
20. Have a history of lack of response to duloxetine or escitalopram at a clinically appropriate dose for a minimum of 4 weeks, or have previously completed or withdrawn from this study or any other study investigating duloxetine or escitalopram.
21. Have any previous diagnosis of bipolar disorder, schizophrenia, or other psychotic disorders.
22. Have DSM-IV-defined history of substance abuse or dependence within the past year, excluding nicotine and caffeine.
23. Have serious or unstable cardiovascular, hepatic, renal, respiratory or hematological illness; symptomatic peripheral vascular disease; or other medical (including unstable hypertension and not clinically euthyroid) or psychological conditions that, in the opinion of the investigator, would compromise participation or be likely to require hospitalization during the course of the study.
24. Have had Electroconvulsive Therapy (ECT) or Transcranial Magnetic Stimulation within the past year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 840 (Actual)
Dates: Start 2008-11; Primary Completion 2010-02 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) Mon-Fri 9AM-5PM Eastern time (UTC/GMT-5 hours, EST), Study Director — Eli Lilly and Company
Locations (60):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Copenhagen, Denmark
- France (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Angoulême
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Arcachon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Dole
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Gujan-Mestras
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Marseille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Montpellier
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Nîmes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Orvault
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Rennes
- Greece (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Athens
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Haidari, Athens
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Thessaloniki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Tripoli
- Hungary (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Balassagyarmat
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Budapest
- Italy (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Chieti
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Foggia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Milan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Modena
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Parma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Pisa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Siena
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Teramo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Terracina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Torino
- Netherlands (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Beek en Donk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Brummen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Brunssum
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Deurne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Heerde
- Romania (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Constanța
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Iași
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Timișoara
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Ljubljana, Slovenia
- Spain (11):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Alcalá de Henares
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Ferrol
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Foios
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Palma de Mallorca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Salamanca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Seville
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal ph, Vigo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Zamora
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Zaragoza
- Sweden (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Gothenburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Halmstad
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Luleå
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Lund
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Malmo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Stockholm
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Sundsvall
- Turkey (Türkiye) (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Ankara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Antakya
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Çapa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Dışkapı
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Izmir
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Şişli

REFERENCES:
- [Derived] Romera I, Perez V, Menchon JM, Schacht A, Papen R, Neuhauser D, Abbar M, Svanborg P, Gilaberte I. Early switch strategy in patients with major depressive disorder: a double-blind, randomized study. J Clin Psychopharmacol. 2012 Aug;32(4):479-86. doi: 10.1097/JCP.0b013e31825d9958. PMID 22722513

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants showing improvement (≥30% baseline score reduction on the HAMD-17) during Period I did not continue to Period II of the study. Qualified participants for Period II were randomized to either Early Intervention Strategy Arm or Delayed Intervention Strategy Arm.
Pre-assignment Details: Baseline demographics and primary and secondary outcomes are reported only for Period II (Double Blind Treatment Strategy). Adverse events (AEs) are reported for Period I (Acute Escitalopram Treatment) and Period II.
Groups:
- Escitalopram (Acute Treatment): Escitalopram 10 milligrams (mg) per day for 4 weeks
- Early Intervention: Duloxetine flexible dose (60 or 120 milligrams [mg] daily) for 12 weeks
- Delayed Intervention: Escitalopram flexible dose (10 to 20 milligrams [mg] daily) for 4 weeks. Then in participants with no-response, switch treatment to duloxetine flexible dose (60 or 120 mg daily) for 8 weeks. In participants with a response continue treatment with escitalopram (10 to 20 milligrams [mg] daily) for 8 weeks.
Period: Lead-in Period I
Arm/Group | Escitalopram (Acute Treatment) | Early Intervention | Delayed Intervention
Started | 840 | 0 | 0
Completed | 566 | 0 | 0
Not Completed | 274 | 0 | 0
Not completed — Adverse Event | 43 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Lost to Follow-up | 19 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 46 | 0 | 0
Not completed — Protocol entry criterion not met | 5 | 0 | 0
Not completed — Randomization criteria not met | 158 | 0 | 0
Period: Double-Blind Period II
Arm/Group | Escitalopram (Acute Treatment) | Early Intervention | Delayed Intervention
Started | 0 | 282 | 284 (At Week 8 - delayed intervention divided by response to treatment (nonresponders or responders).)
Completed | 0 | 226 | 212
Not Completed | 0 | 56 | 72
Not completed — Adverse Event | 0 | 9 | 8
Not completed — Lack of Efficacy | 0 | 7 | 12
Not completed — Lost to Follow-up | 0 | 9 | 9
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 21 | 35
Not completed — Protocol entry criterion not met | 0 | 0 | 1
Not completed — Clinical relapse | 0 | 3 | 0
Not completed — Protocol Violation | 0 | 7 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Early Intervention | Delayed Intervention | Total
Number analyzed (Participants) | 282 | 284 | 566
Age Continuous [Mean (Standard Deviation); unit: years] | 48.3 (13.48) | 47.4 (12.72) | 47.9 (13.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 196 | 197 | 393
  Male | 86 | 87 | 173
Region of Enrollment [Number; unit: participants]
  France | 54 | 54 | 108
  Hungary | 6 | 6 | 12
  Slovenia | 6 | 4 | 10
  Greece | 10 | 10 | 20
  Spain | 71 | 73 | 144
  Turkey | 10 | 10 | 20
  Romania | 18 | 18 | 36
  Denmark | 12 | 14 | 26
  Netherlands | 5 | 4 | 9
  Italy | 19 | 20 | 39
  Sweden | 71 | 71 | 142
Race [Number; unit: participants]
  Black or African American | 2 | 2 | 4
  White | 280 | 282 | 562
Clinical Global Impression-Major Depressive Disorder-Severity (CGI-MDD-S) Score [Mean (Standard Deviation); unit: units on a scale] — Measures severity of illness at the time of assessment compared with start of treatment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill participants.
  units on a scale | 4.6 (0.59) | 4.6 (0.64) | 4.6 (0.62)
Quick Inventory of Depressive Symptomatology-Self Reported (QIDS16SR) Total Score [Mean (Standard Deviation); unit: units on a scale] — A 16-item participant-rated measure of depressive symptomatology. The total score ranges from 0 to 27 with higher scores indicative of greater severity.
  units on a scale | 16.4 (3.82) | 16.7 (3.43) | 16.5 (3.63)
17-item Hamilton Depression Rating Scale (HAMD-17) Total Score [Mean (Standard Deviation); unit: units on a scale] — The 17-item HAMD measures depression severity. Each item was evaluated and scored using either a 5-point scale (e.g. absent, mild, moderate, severe, very severe) or a 3-point scale (e.g. absent, mild, marked). The total score of HAMD-17 may range from 0 (normal) to 52 (severe).
  units on a scale | 24.0 (3.57) | 24.4 (3.83) | 24.2 (3.70)
Visual Analog Scale (VAS) Overall Pain Severity [Mean (Standard Deviation); unit: units on a scale] — VAS for pain consists of 6 questions that assess overall pain, headache, back pain, shoulder pain, pain interference with daily activities, and pain while awake. Participant rates pain on a 10 centimeter (cm) line between two anchors (0= no pain and 10=very severe pain).
  units on a scale | 3.6 (2.76) | 3.8 (2.81) | 3.7 (2.78)
Sheehan Disability Scale (SDS) Total Score [Mean (Standard Deviation); unit: units on a scale] — The SDS is completed by the participant and is used to assess the effect of the participant's symptoms on their work/social/family life. Total scores range from 0 to 30 with higher values indicating greater disruption in the participant's work/social/family life.
  units on a scale | 19.9 (5.12) | 19.9 (5.52) | 19.9 (5.32)
Euro Quality of Life-5 Dimensions Questionnaire (EQ-5D) Score [Mean (Standard Deviation); unit: units on a scale] — EQ-5D: a generic, multidimensional, health-related, quality of life instrument. Participants rate health state in 5 domains: mobility, self-care, usual activities, pain/discomfort, mood. A single score between 1-3 is generated for each domain. Outcome rating on 5 domains is mapped to a single index through an algorithm. Index ranges between 0-1 with higher score indicating better health state perceived by participant. Health State Score: self-rated health on a vertical visual analogue scale measured in centimeters. Best imaginable health state=10 and worst imaginable health state=0.
  units on a scale
    EQ-5D UK Population-based Index Score | 0.40 (0.291) | 0.34 (0.312) | 0.37 (0.303)
    Health State Score | 4.23 (1.873) | 3.86 (1.704) | 4.05 (1.798)
Number of work hours worked per week [Mean (Standard Deviation); unit: hours] | 38.0 (8.30) | 37.2 (9.53) | 37.6 (8.94)
Number of work hours missed in the last 4 weeks [Mean (Standard Deviation); unit: hours] — Only those participants who missed at least 1 hour of work were included: 79 participants in the Early Intervention Strategy group and 93 participants in the Delayed Intervention Strategy group.
  hours | 86.9 (63.09) | 87.5 (66.32) | 87.2 (64.67)
Number of work hours missed due to depression in the last 4 weeks [Mean (Standard Deviation); unit: hours] — Only those participants who missed at least 1 hour of work due to depression were included: 73 participants in the Early Intervention Strategy group and 90 participants in the Delayed Intervention Strategy group.
  hours | 88.8 (64.14) | 88.5 (67.05) | 88.6 (65.56)
Number of visits to primary healthcare provider due to depression in the last 4 weeks [Mean (Standard Deviation); unit: visits] | 1.6 (0.95) | 1.8 (1.10) | 1.7 (1.03)
Number of visits to emergency room or equivalent facility due to depression in the last 4 weeks [Mean (Standard Deviation); unit: visits] | 1.1 (0.27) | 1.1 (0.48) | 1.1 (0.40)
Number of visits to other specialists due to depression in the last 4 weeks [Mean (Standard Deviation); unit: visits] | 2.0 (1.44) | 1.6 (0.98) | 1.8 (1.26)
Has the participant been hospitalized due to depression in the last 4 weeks [Number; unit: participants]
  Yes | 4 | 5 | 9
  No | 277 | 278 | 555
  Unknown | 1 | 0 | 1
  Missing | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Time to Confirmed Response by ≥ 50% Change From Baseline Reduction in the Hamilton Depression Rating Scale-17 Items (HAMD-17)
Description: Time to confirmed response is defined as the time from the day of study randomization (Visit 2) to the date of first observation of confirmed response defined as ≥ 50% baseline score reduction on the HAMD-17 for 2 consecutive visits. The 17-item HAMD measures depression severity. Each item was evaluated and scored using either a 5-point scale, e.g. absent, mild, moderate, severe, very severe) or a 3-point scale (e.g. absent, mild, marked). The total score of HAMD-17 may range from 0 (normal) to 52 (severe).
Time Frame: Week 4 through Week 16
Population: Full Analysis Set
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Early Intervention | Delayed Intervention
Number analyzed (Participants) | 282 | 284
weeks | 6.4 [6.0 to 8.0] | 8.0 [6.4 to 8.6]
Statistical Analysis 1: Comparison: Early Intervention vs Delayed Intervention; Kaplan-Meier Estimates (weeks): analysis of early intervention versus delayed intervention strategies; Test type: Superiority or Other; p = 0.213, Kaplan-Meier Analysis — P-value is for early intervention strategy versus delayed intervention strategy; Kaplan-Meier analysis with Wilcoxon test to compare strategies

2. Primary Outcome: Estimated Probability of Not Reaching Confirmed Response at 12 Weeks Based on the Survival Function for the Time to Confirmed Response
Description: Survival function is estimating the probability of participants not achieving confirmed response after 12 weeks. Confirmed response is defined as >=50% change from baseline reduction in the Hamilton Depression Rating Scale-17 Items (HAMD-17). The 17-item HAMD measures depression severity. Each item was evaluated and scored using either a 5-point scale (e.g. absent, mild, moderate, severe, very severe) or a 3-point scale (e.g. absent, mild, marked). The total score of HAMD-17 may range from 0 (normal) to 52 (severe).
Time Frame: Week 4 through Week 16
Population: Full Analysis Population
Measure: Mean (95% Confidence Interval); unit: estimated probability (percent)
Arm/Group | Early Intervention | Delayed Intervention
Number analyzed (Participants) | 282 | 284
estimated probability (percent) | 28 [22 to 34] | 26 [20 to 32]
Statistical Analysis 1: Comparison: Early Intervention vs Delayed Intervention; Survival function estimated over a 12 week period (Week 4 through Week 16): analysis of early intervention versus delayed intervention strategies; Test type: Superiority or Other; p = 0.653, Kaplan Meier analysis — P-value is for comparison of early intervention versus delayed intervention as a function of survival rate over a 12 week period (Week 4 through Week 16); P-value for comparison of rates is based on normal approximation using Greenwood's estimation for standard error; survival rate difference = 0.02, 95% CI 2-sided [-0.06 to 0.10]

3. Secondary Outcome: Time to Confirmed Response as Defined by ≥ 50% Reduction From Baseline Reduction in the 16-Item Quick Inventory of Depressive Symptomatology Self Report (QIDS16SR) That is Reported for Two Consecutive Visits
Description: Time to confirmed response is defined as the time from the day of study randomization (Visit 2) to the date of first observation of confirmed response. QIDS16SR is a 16-item participant-rated measure of depressive symptomatology. The total score ranges from 0 to 27 with higher scores indicative of greater severity.
Time Frame: Week 4 through Week 16
Population: Full Analysis Population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Early Intervention | Delayed Intervention
Number analyzed (Participants) | 282 | 284
weeks | 6.0 [5.0 to 8.0] | 6.9 [5.3 to 8.0]
Statistical Analysis 1: Comparison: Early Intervention vs Delayed Intervention; Analysis of early intervention strategy versus delayed intervention strategy; Test type: Superiority or Other; p = 0.947, Kaplan Meier analysis — P-value is for early intervention strategy versus delayed intervention strategy; Kaplan-Meier analysis with Wilcoxon test to compare strategies

4. Secondary Outcome: Time to Confirmed Remission as Defined by a 16-Item Quick Inventory of Depressive Symptomatology Self Report (QIDS16SR) Score of ≤ 5 That is Maintained for Two Consecutive Visits.
Description: Time to confirmed remission is defined as the time from the day of study randomization (Visit 2) to the date of first observation of confirmed remission. A 16-item participant-rated measure of depressive symptomatology. The total score ranges from 0 to 27 with higher scores indicative of greater severity.
Time Frame: Week 4 through Week 16
Population: Full Analysis Population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Early Intervention | Delayed Intervention
Number analyzed (Participants) | 280 | 284
weeks | NA [12.3 to NA] — It could not be estimated due to the low number of events. | NA [12.3 to NA] — It could not be estimated due to the low number of events.
Statistical Analysis 1: Comparison: Early Intervention vs Delayed Intervention; Analysis of early intervention strategy versus delayed intervention strategy; Test type: Superiority or Other; p = 0.597, Kaplan-Meier analysis — P-value is for early intervention versus delayed intervention strategies; Kaplan-Meier analysis with Wilcoxon test to compare strategies

5. Secondary Outcome: Clinical Global Impressions of Severity (CGI-S) Scale
Description: Measures severity of illness at the time of assessment compared with start of treatment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill participants).
Time Frame: Baseline, Week 4, Week 6, Week 8, Week 10, Week 12, Week 14, Week 16
Population: Full Analysis Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Early Intervention | Delayed Intervention
Number analyzed (Participants) | 282 | 284
units on a scale
  Baseline (n=282, 284) | 4.6 (0.59) | 4.6 (0.64)
  Week 4 (n=281, 284) | 4.3 (0.61) | 4.3 (0.66)
  Week 6 (n=271, 277) | 3.6 (0.88) | 3.7 (0.97)
  Week 8 (n=254, 254) | 3.2 (1.11) | 3.3 (1.15)
  Week 10 (n=231, 236) | 2.8 (1.17) | 2.9 (1.22)
  Week 12 (n=203, 214) | 2.6 (1.21) | 2.7 (1.20)
  Week 14 (n=184, 194) | 2.4 (1.13) | 2.5 (1.17)
  Week 16 (n=178, 182) | 2.2 (1.09) | 2.2 (1.11)
Statistical Analysis 1: Comparison: Early Intervention vs Delayed Intervention; Repeated Measurements Analysis: Early Intervention versus Delayed Intervention Strategy at Week 6; Test type: Superiority or Other; p = 0.624, Mixed Models Analysis — P-value for Week 6: Analysis of early versus delayed intervention strategies LS Mean/Estimate; Mixed models repeated measures with fixed effects for strategy, country, visit, strategy-by-visit interaction, baseline score and baseline-by visit; LS Mean = -0.04, 95% CI 2-sided [-0.22 to 0.13], Standard Error of Mean 0.09
Statistical Analysis 2: Comparison: Early Intervention vs Delayed Intervention; Repeated Measurements Analysis: Early Intervention versus Delayed Intervention Strategy at Week 8; Test type: Superiority or Other; p = 0.208, Mixed Models Analysis — P-value for Week 8: Analysis of early versus delayed intervention strategies LS Mean/Estimate; Mixed Models repeated measures with fixed effects for strategy, country, visit, strategy-by-visit interaction, baseline score and baseline-by-visit; LS Mean = -0.11, 95% CI 2-sided [-0.29 to 0.06], Standard Error of Mean 0.09
Statistical Analysis 3: Comparison: Early Intervention vs Delayed Intervention; Repeated Measurements Analysis: Early Intervention versus Delayed Intervention Strategy at Week 10; Test type: Superiority or Other; p = 0.044, Mixed Models Analysis — P-value for Week 10: Analysis of early versus delayed intervention strategies LS Mean/Estimate; [statistical method as in outcome 5, analysis 2]; LS Mean = -0.19, 95% CI 2-sided [-0.37 to -0.00], Standard Error of Mean 0.09
Statistical Analysis 4: Comparison: Early Intervention vs Delayed Intervention; Repeated Measurements Analysis: Early Intervention versus Delayed Intervention Strategy at Week 12; Test type: Superiority or Other; p = 0.086, Mixed Models Analysis — P-value for Week 12: Analysis of early versus delayed intervention strategies LS Mean/Estimate; Mixed models repeated measures with fixed effects for strategy, country, visit, strategy-by-visit interactions, baseline score and baseline-by-visit; LS Mean = -0.16, 95% CI 2-sided [-0.35 to 0.02], Standard Error of Mean 0.10
Statistical Analysis 5: Comparison: Early Intervention vs Delayed Intervention; Repeated Measurements Analysis: Early Intervention versus Delayed Intervention Strategy at Week 14; Test type: Superiority or Other; p = 0.181, Mixed Models Analysis — P-value for Week 14: Analysis of early versus delayed intervention strategies LS Mean/Estimate; [statistical method as in outcome 5, analysis 2]; LS Mean = -0.13, 95% CI 2-sided [-0.33 to 0.06], Standard Error of Mean 0.10
Statistical Analysis 6: Comparison: Early Intervention vs Delayed Intervention; Repeated Measurements Analysis: Early Intervention versus Delayed Intervention Strategy at Week 16; Test type: Superiority or Other; p = 0.994, Mixed Models Analysis — P-value for Week 16: Analysis of early versus delayed intervention strategies LS Mean/Estimate; [statistical method as in outcome 5, analysis 2]; LS Mean = 0.00, 95% CI 2-sided [-0.20 to 0.20], Standard Error of Mean 0.10

6. Secondary Outcome: Visual Analog Scale (VAS) - Overall Pain Severity
Description: VAS for pain consists of 6 questions that assess overall pain, headache, back pain, shoulder pain, pain interference with daily activities, and pain while awake. Participant rates pain on a 10 centimeter (cm) line between two anchors (0= no pain and 10=very severe pain).
Time Frame: Baseline, Week 4, Week 6, Week 8, Week 10, Week 12, Week 14, Week 16
Population: Full Analysis Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Early Intervention | Delayed Intervention
Number analyzed (Participants) | 282 | 284
units on a scale
  Baseline (n=282, 284) | 3.6 (2.76) | 3.8 (2.81)
  Week 4 (n=281, 283) | 3.0 (2.54) | 3.5 (2.77)
  Week 6 (n=270, 271) | 2.6 (2.41) | 3.3 (2.85)
  Week 8 (n=245, 241) | 2.4 (2.53) | 3.0 (2.70)
  Week 10 (n=207, 204) | 2.4 (2.48) | 2.7 (2.60)
  Week 12 (n=170, 181) | 2.1 (2.42) | 2.6 (2.66)
  Week 14 (n=151, 152) | 2.0 (2.35) | 2.5 (2.54)
  Week 16 (n=143, 152) | 2.0 (2.32) | 2.3 (2.55)
Statistical Analysis 1: Comparison: Early Intervention vs Delayed Intervention; Repeated Measurements Analysis: Early Intervention versus Delayed Intervention Strategy at Week 6; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis — P-value for Week 6: Analysis of early versus delayed intervention strategies LS Mean/Estimate; [statistical method as in outcome 5, analysis 1]; LS Mean = -0.62, 95% CI 2-sided [-0.98 to -0.25], Standard Error of Mean 0.19
Statistical Analysis 2: Comparison: Early Intervention vs Delayed Intervention; Repeated Measurements Analysis: Early Intervention versus Delayed Intervention Strategy at Week 8; Test type: Superiority or Other; p = 0.010, Mixed Models Analysis — P-value for Week 8: Analysis of early versus delayed intervention strategies LS Mean/Estimate; [statistical method as in outcome 5, analysis 2]; LS Mean = -0.50, 95% CI 2-sided [-0.87 to -0.12], Standard Error of Mean 0.19
Statistical Analysis 3: Comparison: Early Intervention vs Delayed Intervention; Repeated Measurements Analysis: Early Intervention versus Delayed Intervention Strategy at Week 10; Test type: Superiority or Other; p = 0.445, Mixed Models Analysis — P-value for Week 10: analysis of early versus delayed intervention strategies LS Mean/Estimate; [statistical method as in outcome 5, analysis 2]; LS Mean = -0.15, 95% CI 2-sided [-0.55 to 0.24], Standard Error of Mean 0.20
Statistical Analysis 4: Comparison: Early Intervention vs Delayed Intervention; Repeated Measurements Analysis: Early Intervention versus Delayed Intervention Strategy at Week 12; Test type: Superiority or Other; p = 0.169, Mixed Models Analysis — P-value for Week 12: Analysis of early versus delayed intervention strategies LS Mean/Estimate; [statistical method as in outcome 5, analysis 2]; LS Mean = -0.29, 95% CI 2-sided [-0.71 to 0.12], Standard Error of Mean 0.21
Statistical Analysis 5: Comparison: Early Intervention vs Delayed Intervention; Repeated Measurements Analysis: Early Intervention versus Delayed Intervention Strategy at Week 14; Test type: Superiority or Other; p = 0.393, Mixed Models Analysis — P-value for Week 14: Analysis of early versus delayed intervention strategies LS Mean/Estimate; [statistical method as in outcome 5, analysis 2]; LS Mean = -0.19, 95% CI 2-sided [-0.63 to 0.25], Standard Error of Mean 0.23
Statistical Analysis 6: Comparison: Early Intervention vs Delayed Intervention; Repeated Measurements Analysis: Early Intervention versus Delayed Intervention Strategy at Week 16; Test type: Superiority or Other; p = 0.510, Mixed Models Analysis — P-value for Week 16: Analysis of early versus delayed intervention strategies LS Mean/Estimate; Mixed models repeated measures with fixed effects for strategy, country, visit, strategy-by-visit interaction, baseline scores and baseline-by-visit; LS Mean = -0.15, 95% CI 2-sided [-0.61 to 0.30], Standard Error of Mean 0.23

7. Secondary Outcome: Euro Quality of Life Questionnaire-5 Dimensions (EQ-5D) Scale - Health State Score
Description: The EQ-5D Health State Score is self-rated health on a vertical, visual analogue scale measured in centimeters (cm) and reported as units on a scale. Best imaginable health state = 10 cm and worst imaginable health state = 0 cm.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 16
Population: Full Analysis Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Early Intervention | Delayed Intervention
Number analyzed (Participants) | 282 | 283
units on a scale
  Baseline (n=281, 283) | 4.2 (1.87) | 3.9 (1.70)
  Week 4 (n=282, 280) | 4.9 (1.76) | 4.5 (1.62)
  Week 8 (n=244, 237) | 5.7 (1.88) | 5.4 (1.94)
  Week 12 (n=169, 177) | 5.9 (1.96) | 5.8 (1.98)
  Week 16 (n=142, 153) | 6.5 (1.90) | 6.5 (1.94)
Statistical Analysis 1: Comparison: Early Intervention vs Delayed Intervention; Repeated Measurements Analysis: Early Intervention versus Delayed Intervention Strategy at Week 8; Test type: Superiority or Other; p = 0.401, Mixed Models Analysis — P-value for Week 8: Analysis of early intervention versus delayed intervention strategies LS Mean/Estimate; [statistical method as in outcome 5, analysis 2]; LS Mean = 0.14, 95% CI 2-sided [-0.19 to 0.47], Standard Error of Mean 0.17
Statistical Analysis 2: Comparison: Early Intervention vs Delayed Intervention; Repeated Measurements Analysis: Early Intervention versus Delayed Intervention Strategy at Week 12; Test type: Superiority or Other; p = 0.618, Mixed Models Analysis — P-value for Week 12: Analysis of early intervention versus delayed intervention strategies LS Mean/Estimate; [statistical method as in outcome 5, analysis 2]; LS Mean = 0.09, 95% CI 2-sided [-0.27 to 0.46], Standard Error of Mean 0.19
Statistical Analysis 3: Comparison: Early Intervention vs Delayed Intervention; Repeated Measurements Analysis: Early Intervention versus Delayed Intervention Strategy at Week 16; Test type: Superiority or Other; p = 0.856, Mixed Models Analysis — P-value for Week 16: Analysis of early intervention versus delayed intervention strategies LS Mean/Estimate; [statistical method as in outcome 5, analysis 2]; LS Mean = -0.04, 95% CI 2-sided [-0.43 to 0.36], Standard Error of Mean 0.20

8. Secondary Outcome: Euro Quality of Life Questionnaire-5 Dimensions (EQ-5D) Scale - United Kingdom (UK) Population Based Index Score
Description: The EQ-5D is a generic, multidimensional, health-related, quality of life instrument. The profile allows participants to rate their health state in 5 health domains: mobility, self-care, usual activities, pain/discomfort, and mood. A single score between 1 and 3 is generated for each domain. For each participant, the outcome rating on the 5 domains will be mapped to a single index through an algorithm. The index ranges between 0 and 1, with the higher score indicating a better health state perceived by the participant.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 16
Population: Full Analysis Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Early Intervention | Delayed Intervention
Number analyzed (Participants) | 279 | 282
units on a scale
  Baseline (n=279, 282) | 0.4 (0.29) | 0.3 (0.31)
  Week 4 (n=279, 282) | 0.5 (0.30) | 0.5 (0.32)
  Week 8 (n=244, 238) | 0.7 (0.25) | 0.6 (0.30)
  Week 12 (n=168, 178) | 0.7 (0.22) | 0.6 (0.28)
  Week 16 (n=143, 153) | 0.7 (0.24) | 0.7 (0.24)
Statistical Analysis 1: Comparison: Early Intervention vs Delayed Intervention; Repeated Measurements Analysis: Early Intervention versus Delayed Intervention Strategy at Week 8; Test type: Superiority or Other; p = 0.021, Mixed Models Analysis — P-value for Week 8: Analysis of early versus delayed intervention LS Mean/Estimate; [statistical method as in outcome 5, analysis 2]; LS Mean = -0.05, 95% CI 2-sided [-0.10 to -0.01], Standard Error of Mean 0.02
Statistical Analysis 2: Comparison: Early Intervention vs Delayed Intervention; Repeated Measurements Analysis: Early Intervention versus Delayed Intervention Strategy at Week 12; Test type: Superiority or Other; p = 0.071, Mixed Models Analysis — P-value for Week 12: Analysis of early versus delayed intervention strategies LS Mean/Estimate; [statistical method as in outcome 5, analysis 2]; LS Mean = -0.04, 95% CI 2-sided [-0.09 to 0.00], Standard Error of Mean 0.02
Statistical Analysis 3: Comparison: Early Intervention vs Delayed Intervention; Repeated Measurements Analysis: Early Intervention versus Delayed Intervention Strategy at Week 16; Test type: Superiority or Other; p = 0.792, Mixed Models Analysis — P-value for Week 16: Analysis of early versus delayed intervention strategies LS Mean/Estimate; [statistical method as in outcome 5, analysis 2]; LS Mean = 0.01, 95% CI 2-sided [-0.05 to 0.06], Standard Error of Mean 0.03

9. Secondary Outcome: Sheehan Disability Scale (SDS) Normal Functioning Total Score
Description: The SDS is completed by the participant and is used to assess the effect of the participant's symptoms on their work/social/family life. Total scores range from 0 to 30 with higher values indicating greater disruption in the participant's work/social/family life.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 16
Population: Full Analysis Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Early Intervention | Delayed Intervention
Number analyzed (Participants) | 216 | 217
units on a scale
  Baseline (n=216, 217) | 19.9 (5.12) | 19.9 (5.52)
  Week 4 (n=215, 215) | 16.9 (6.36) | 17.5 (6.11)
  Week 8 (n=186, 188) | 13.5 (6.50) | 14.0 (6.79)
  Week 12 (n=140, 144) | 12.1 (6.84) | 13.2 (7.51)
  Week 16 (n=113, 121) | 10.3 (7.27) | 10.2 (6.97)
Statistical Analysis 1: Comparison: Early Intervention vs Delayed Intervention; Repeated Measurements Analysis: Early Intervention versus Delayed Intervention Strategy at Week 8; Test type: Superiority or Other; p = 0.597, Mixed Models Analysis — P-value for Week 8: Analysis of early versus delayed intervention strategies LS Mean/Estimate; [statistical method as in outcome 5, analysis 2]; LS Mean = -0.37, 95% CI 2-sided [-1.74 to 1.00], Standard Error of Mean 0.70
Statistical Analysis 2: Comparison: Early Intervention vs Delayed Intervention; Repeated Measurements Analysis: Early Intervention versus Delayed Intervention Strategy at Week 12; Test type: Superiority or Other; p = 0.360, Mixed Models Analysis — P-value for Week 12: Analysis for early versus delayed intervention strategies LS Mean/Estimate; [statistical method as in outcome 5, analysis 2]; LS Mean = -0.68, 95% CI 2-sided [-2.13 to 0.78], Standard Error of Mean 0.74
Statistical Analysis 3: Comparison: Early Intervention vs Delayed Intervention; Repeated Measurements Analysis: Early Intervention versus Delayed Intervention Strategy at Week 16; Test type: Superiority or Other; p = 0.937, Mixed Models Analysis — P-value for Week 16: Analysis for early versus delayed intervention strategies LS Mean/Estimate; [statistical method as in outcome 5, analysis 2]; LS Mean = 0.06, 95% CI 2-sided [-1.52 to 1.65], Standard Error of Mean 0.81

10. Primary Outcome: Time to Confirmed Remission by a Hamilton Depression Rating Scale-17 Items (HAMD-17) Score of ≤ 7 That is Maintained for Two Consecutive Visits
Description: Time to confirmed remission is defined as the time from the day of study randomization (Visit 2) to the date of first observation of confirmed remission defined as a score on the HAMD-17 of ≤ 7 for 2 consecutive visits. The 17-item HAMD measures depression severity. Each item was evaluated and scored using either a 5-point scale (e.g. absent, mild, moderate, severe, very severe) or a 3-point scale (e.g. absent, mild, marked). The total score of HAMD-17 may range from 0 (normal) to 52 (severe).
Time Frame: Week 4 through Week 16
Population: Full Analysis Population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Early Intervention | Delayed Intervention
Number analyzed (Participants) | 282 | 284
weeks | 12.9 [11.0 to NA] — No maximum value was reported for the 95% confidence interval. It was not reported as it could not be estimated due to the low number of events. | NA [12.3 to NA] — 50% remission (median) could not be estimated for delayed intervention arm due to the low number of events.
Statistical Analysis 1: Comparison: Early Intervention vs Delayed Intervention; Kaplan-Meier estimates (weeks): analysis of early intervention versus delayed intervention strategies; Test type: Superiority or Other; p = 0.075, Kaplan-Meier analysis — P-value is for early intervention strategy versus delayed intervention strategy; Kaplan-Meier analysis with Wilcoxon test to compare strategies

11. Primary Outcome: Estimated Probability of Not Reaching Confirmed Remission at 12 Weeks Based on the Survival Function for the Time to Confirmed Remission
Description: Survival function is estimating the probability of participants not achieving confirmed remission. Confirmed remission is defined as a Hamilton Depression Rating Scale-17 Items (HAMD-17) Score of ≤ 7 that is maintained for two consecutive visits. The 17-item HAMD measures depression severity. Each item was evaluated and scored using either a 5-point scale (e.g. absent, mild, moderate, severe, very severe) or a 3-point scale (e.g. absent, mild, marked). The total score of HAMD-17 may range from 0 (normal) to 52 (severe).
Time Frame: Week 4 through Week 16
Population: Full Analysis Population
Measure: Mean (95% Confidence Interval); unit: estimated probability (percent)
Arm/Group | Early Intervention | Delayed Intervention
Number analyzed (Participants) | 282 | 284
estimated probability (percent) | 52 [46 to 58] | 59 [53 to 66]
Statistical Analysis 1: Comparison: Early Intervention vs Delayed Intervention; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.116, Kaplan-Meier analysis — [p-value comment as in outcome 2, analysis 1]; P-value for comparison of rates is based on normal approximation using Greenwood's estimation for standard error; Survival rate difference = -0.07, 95% CI 2-sided [-0.16 to 0.02]

12. Secondary Outcome: Resource Utilisation - Number of Hours Worked Per Week
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 16
Population: Full Analysis Population, which included all randomized participants with at least 1 post-randomization assessment available after Week 4. For efficacy analyses, participants were included in the analysis if they had a baseline and a post-baseline (after Week 4) value of the variable in question.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Early Intervention | Delayed Intervention
Number analyzed (Participants) | 282 | 284
Hours
  Week 4 (n=153, 159) | 37.7 (11.61) | 38.6 (13.33)
  Week 8 (n=136, 141) | 37.9 (9.08) | 37.7 (8.42)
  Week 12 (n=119, 115) | 37.7 (7.40) | 38.1 (13.72)
  Week 16 (n=96, 96) | 37.2 (7.80) | 38.0 (14.74)

13. Secondary Outcome: Resource Utilisation - Number of Work Hours Missed in the Last 4 Weeks
Description: Only those participants who missed at least 1 hour of work were included.
Time Frame: Week 4, Week 8, Week 12, Week 16
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Early Intervention | Delayed Intervention
Number analyzed (Participants) | 282 | 284
Hours
  Week 4 (n=73, 89) | 88.6 (64.30) | 95.0 (67.40)
  Week 8 (n=54, 67) | 92.5 (66.12) | 102.3 (69.38)
  Week 12 (n=38, 56) | 85.0 (65.73) | 104.5 (68.72)
  Week 16 (n=25, 39) | 91.5 (63.49) | 126.4 (63.64)

14. Secondary Outcome: Resource Utilisation - Number of Work Hours Missed Due to Depression in the Last 4 Weeks
Description: Only those participants who missed at least 1 hour of work due to depression were included.
Time Frame: Week 4, Week 8, Week 12, Week 16
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Early Intervention | Delayed Intervention
Number analyzed (Participants) | 282 | 284
Hours
  Week 4 (n=70, 86) | 90.6 (64.98) | 95.1 (67.90)
  Week 8 (n=47, 61) | 98.5 (65.34) | 109.7 (68.08)
  Week 12 (n=31, 52) | 98.7 (64.32) | 111.4 (66.42)
  Week 16 (n=24, 38) | 91.9 (64.99) | 126.0 (63.40)

15. Secondary Outcome: Resource Utilisation - Number of Visits to Primary Healthcare Provider Due to Depression in the Last 4 Weeks
Time Frame: Week 4, Week 8, Week 12, Week 16
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Visits
Arm/Group | Early Intervention | Delayed Intervention
Number analyzed (Participants) | 282 | 284
Visits
  Week 4 (n=36, 55) | 1.5 (1.00) | 1.6 (1.04)
  Week 8 (n=14, 22) | 1.1 (0.27) | 1.7 (1.13)
  Week 12 (n=8, 12) | 1.3 (0.46) | 1.6 (1.00)
  Week 16 (n=4, 7) | 2.0 (2.00) | 1.6 (1.13)

16. Secondary Outcome: Resource Utilisation - Number of Visits to Other Specialists Due to Depression in the Last 4 Weeks
Time Frame: Week 4, Week 8, Week 12, Week 16
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Visits
Arm/Group | Early Intervention | Delayed Intervention
Number analyzed (Participants) | 282 | 284
Visits
  Week 4 (n=25, 16) | 2.2 (2.05) | 1.7 (0.87)
  Week 8 (n=8, 8) | 1.6 (0.74) | 1.9 (1.13)
  Week 12 (n=3, 2) | 1.7 (1.15) | 1.0 (0.00)
  Week 16 (n=2, 1) | 2.0 (0.00) | 3.0 (NA) — n=1 participant; therefore SD could not be calculated.

17. Secondary Outcome: Resource Utilisation - Has the Participant Been Hospitalized Due to Depression in the Last 4 Weeks - Number of Participants With a Yes Response
Time Frame: Week 4, Week 8, Week 12, Week 16
Population: Full Analysis Population
Measure: Number; unit: participants
Arm/Group | Early Intervention | Delayed Intervention
Number analyzed (Participants) | 282 | 284
participants
  Week 4 | 1 | 0
  Week 8 | 0 | 0
  Week 12 | 0 | 0
  Week 16 | 0 | 0

18. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: The list of AEs is located in the Reported Adverse Event module.
Time Frame: Baseline through Week 16
Population: Full Analysis Population
Measure: Number; unit: participants
Arm/Group | Early Intervention | Delayed Intervention
Number analyzed (Participants) | 282 | 284
participants
  Number of participants with adverse events | 112 | 101
  Number of participants with serious adverse events | 8 | 4

ADVERSE EVENTS:
Description: Adverse events section reports events for participants in Period I (840) and Period II (282 early intervention, 284 delayed intervention). During Period II (Week 8), delayed intervention participants were subdivided by response to treatment (165 non-responders, 83 responders) and adverse events experienced by these participants are reported here.
Groups:
- Escitalopram (Acute Treatment): Escitalopram 10 mg per day for 4 weeks (one 10 mg-capsule)
- Delayed Intervention (Double Blind): Escitalopram 10 to 20 mg per day for 4 weeks (one or two 10 mg capsule[s]). Then, non-responders switched to duloxetine 60 or 120 mg per day for 8 weeks, and responders continued on escitalopram 10 to 20 mg per day for 8 weeks.
- Early Intervention (Double Blind): Duloxetine flexible dose (60 or 120 milligram [mg] daily) for 12 weeks.
- Delayed Intervention Responders: Escitalopram 10 to 20 mg per day for 8 weeks.
- Delayed Intervention Non-Responders: Duloxetine 60 or 120 mg per day for 8 weeks.
Arm/Group | Escitalopram (Acute Treatment) | Delayed Intervention (Double Blind) | Early Intervention (Double Blind) | Delayed Intervention Responders | Delayed Intervention Non-Responders
Serious Adverse Events (participants affected / at risk) | 4/840 | 4/284 | 8/282 | 1/83 | 1/165
Other Adverse Events (participants affected / at risk) | 245/840 | 99/284 | 110/282 | 33/83 | 60/165
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Escitalopram (Acute Treatment) (N=840) | Delayed Intervention (Double Blind) (N=284) | Early Intervention (Double Blind) (N=282) | Delayed Intervention Responders (N=83) | Delayed Intervention Non-Responders (N=165)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug exposure during pregnancy (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intraocular pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abnormal behaviour (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Escitalopram (Acute Treatment) (N=840) | Delayed Intervention (Double Blind) (N=284) | Early Intervention (Double Blind) (N=282) | Delayed Intervention Responders (N=83) | Delayed Intervention Non-Responders (N=165)
Abdominal pain upper (Gastrointestinal disorders) | 10 (10) | 4 (4) | 1 (1) | 1 (1) | 3 (3)
Constipation (Gastrointestinal disorders) | 14 (14) | 2 (2) | 7 (7) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 16 (16) | 6 (6) | 7 (7) | 1 (1) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 26 (28) | 3 (3) | 10 (10) | 2 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastric disorder (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 63 (63) | 5 (5) | 14 (14) | 1 (1) | 4 (4)
Vomiting (Gastrointestinal disorders) | 5 (5) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 7 (7) | 7 (7) | 6 (6) | 4 (4) | 2 (2)
Malaise (General disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Seasonal allergy (Immune system disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 3 (3) | 3 (3) | 5 (5) | 2 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 10 (10) | 12 (13) | 5 (5) | 3 (4) | 9 (9)
Biopsy uterus (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood pressure diastolic decreased (Investigations) | 3 (3) | 2 (2) | 5 (5) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 4 (4) | 4 (4) | 1 (1) | 2 (2) | 2 (2)
Weight increased (Investigations) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) | 1 (1) | 1 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 5 (5) | 2 (2) | 1 (1) | 4 (4)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 15 (15) | 5 (5) | 11 (11) | 3 (3) | 2 (2)
Headache (Nervous system disorders) | 43 (51) | 24 (28) | 22 (43) | 5 (7) | 17 (19)
Somnolence (Nervous system disorders) | 6 (6) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Tension headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 7 (7) | 2 (2) | 3 (3) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 10 (10) | 3 (4) | 2 (2) | 1 (1) | 2 (3)
Insomnia (Psychiatric disorders) | 10 (10) | 4 (4) | 6 (9) | 1 (1) | 3 (3)
Loss of libido (Psychiatric disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Ejaculation delayed (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 20 (20) | 6 (6) | 12 (12) | 5 (5) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
Diastolic hypertension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 2 (2) | 0 (0) | 5 (5) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 19 (19) | 2 (2) | 5 (5) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 5 (5) | 2 (3) | 1 (1) | 1 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days